CLINICAL TRIAL: NCT04827420
Title: Mi QUIT CARE (Mile Square QUIT Community-Access-Referral-Expansion)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alicia Matthews, Professor, Columbia University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-0532; 1UG3HL151302-01 (NIH); 4UH3HL151302-04 (NIH)
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Tobacco Use Cessation
Keywords: Smoking cessation; Federally qualified health care centers; Tobacco quitlines; Implementation Science
MeSH Terms: conditions — Tobacco Use Cessation; Smoking Cessation

STUDY DESIGN:
Intervention Model Description: We are proposing a hybrid type 3 implementation study design (Figure 1) to test the feasibility of delivering tobacco cessation (Advise and Refer components of "AAR") via MyChart/patient portal messaging. We will assess three message types by randomly assigning patients enrolled in MyChart to receive one of three messages - Arm 1: (Choice message + Facilitated referral), Arm 2: (Quit-only + Facilitated referral), or Arm 3 (ITQL Information-only + self-referral). If the patient opts-in to be referred to the quitline, the ITQL will offer an initial intake session to establish treatment goals and then their standard treatment plan.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MiQuit Care (Experimental): Intervention arm: Advise to quit + automatic linkage to quitline + patient navigation
  Interventions: Behavioral: Mi Quit Care
- Enhanced Standard of Care (Active Comparator): Active Comparator: Advise to quit + written self-help materials
  Interventions: Behavioral: Mi Quit Care

INTERVENTIONS:
Behavioral: Mi Quit Care — Demonstrating the feasibility, effectiveness, and cost-effectiveness of electronically delivered smoking cessation interventions via patient portals in Federally Qualified Health Care (FQHC) settings has the potential for wide-spread dissemination and significant public health impact. on patient populations with demonstrated high rates of smoking.

SUMMARY:
The over-arching research question is: Does message (Advise) and referral approach (Refer) influence a patient's willingness to "opt-in" to receive a call from an Illinois Tobacco Quitline (ITQL) smoking cessation coach in patients at MSHC.

Primary UH3 study aim: Compare the effect of the portal-delivered Choice message (Arm 1) to the Information-only message (Arm 3) on linkage to the Illinois Tobacco Quitline (i.e., spoke to a Quitline coach).

Secondary UH3 aims are to:

Examine the reach of the patient portal for delivering "Advise" and "Refer" at 4 weeks. Reach is defined as a patient opening the portal-delivered provider message across all three Arms.

Compare the effect of the Quit message (Quit, Arm 2) to Information-only (Arm 3) on linkage to ITQL.

Compare the effect of the Facilitated-referral messages (opt-in link in the message: Arm 1 & 2) vs. Self-referral (Information-only, Arm 3) on linkage to the ITQL (speaking to an ITQL coach) at four weeks.

Compare the effect of the portal-message content of the Choice message (Arm 1) vs. the Quit message (Arm 2) on linkage acceptance (opting in to be called by the ITQL) at 4 weeks.

Compare the effectiveness of re-engagement message 1 to message 2 for linkage to the ITQL among patients who opted-in to an ITQL call but who were not reached after 3 attempts.

Evaluate the cost-effectiveness of using a patient portal to advise patients to change their smoking behavior and refer them to the ITQL. We will compare the costs associated with our project to the costs associated with advising and referring patients during clinical appointments.

DETAILED DESCRIPTION:
Mi Quit Care is a multi-site study with principal investigators at UIC and Columbia University. Dr. Rachel Caskey is the UIC PI who will oversee all research activities held at UIC and Mile Square Health Center. This includes data collection, intervention delivery, collaboration with community partner, Illinois Tobacco Quitline and Mile Square. Dr. Matthews is the Columbia University PI and who has emirates status at UIC. Their involvement in the study includes the following: involved in meetings, problem solving barriers, monitoring safe and secure data transfer, data analysis and interpretation for de-identified data, dissemination of study results, preparing for future grants, mentoring students, and lead manuscript development. UIC is the grant holder and the IRB of record. A subcontract is in place for Columbia University's involvement (Reference Award 114805). The collaboration of both university in conjunction with the Illinois Tobacco Quitline will create a study to address a simplified version of Ask, Advise, Refer (AAR).

Smoking is the leading preventable cause of death in the U.S. To address this pervasive health risk behavior, all federally qualified health care centers (FQHC) are mandated to provide smoking cessation treatment to all patients who smoke. In 2000, the U.S. Public Health Service clinical practice guideline, Treating Tobacco Use and Dependence, recommended that providers identify and document patients' tobacco use status and treat tobacco users via the "5As" framework (Ask-Advise-Assess-Assist-Arrange). Although effective, the 5As model is time-consuming and challenging to implement. A simplified version (Ask, Advise, Refer, AAR) was developed that resulted in increased patient engagement with recommended treatment approaches such as tobacco quitlines when implemented in clinical settings. Nevertheless, providers continue to experience barriers to the consistent delivery of smoking cessation treatments due to lack of knowledge about appropriate treatments, time constraints, the false belief that most patients are not interested in quitting, and concerns that addressing smoking cessation with their patients may damage the patient provider relationship. Given the high rates of smoking among patients at FQHC settings and the federal mandate to address smoking cessation among all smokers, additional efforts are needed to improve the delivery of care for high-risk and vulnerable populations of smokers.

Implementation science and research approaches are extremely valuable for addressing the unacceptable gap between the demonstration of effective treatments such as "AAR" and barriers to adoption in clinical practice settings. In preparation for a larger Type 3 hybrid implementation-effectiveness study, the purpose of this feasibility study is to evaluate implementation approaches for improving the delivery of the current standard of care smoking cessation treatments (AAR) at Mile Square Health Center (MSHC). The primary goal of the study is to test strategies that can improve the consistent delivery of current standard of care tobacco reduction activities used by providers at MSHC. The study will utilize retrospective chart reviews to identify patients who smoke and extend the current standard of care activities related to smoking cessation treatment. The current MSHC standard of care activities related to smoking cessation treatment include: 1) delivery of "Ask, Advise" by clinic staff and providers then 2) provider "Referral" of patients to the Illinois Tobacco Quitline (ITQL) for free or low-cost smoking cessation treatment. Implementation strategies from the feasibility trial will be integrated into the larger Type 3 implementation-effectiveness randomized controlled trial.

The primary innovation of this study is the use of the Epic linked UI Health Patient Portal platform (MyChart) to deliver the smoking cessation treatment to MSHC patients. This form of delivery is an extension of the current standard of care given at MSHC. Patient portals are secure online websites that give patients convenient, 24-hour access to personal health information from anywhere with an Internet connection. Patient portals have demonstrated benefits for improving patient provider communication, management of chronic health conditions, and patient satisfaction. Patient portals are increasingly being used to deliver health promotion interventions, with positive benefits. However, to our knowledge, no prior projects have examined the use of patient portals to standardize the delivery of referrals for smoking cessation treatment to patients who smoke. This study extends the standard of care to the patient portal. MSHC providers acknowledge inconsistently following the standard of care during clinic visits, and thus, this study proposes to deliver these messages (advise and refer) via the patient portal to increase consistency in message delivery and improve patient access to the standard of care. Because the patient portal was established so providers could communicate with their patients about their health needs, the proposed research is consistent with this goal by using the portal to deliver the same messages. That said, sending provider messages via the patient portal is not the standard of care and instead represents research to convey the messages using a more accessible and reliable approach.

Ask is completed as part of routine care and captured in the medical record. We will use the data documented from "Ask" to identify smokers to send our messages (Advise and Refer). We will test strategies to revise and extend the delivery of the Advise and Refer components of "AAR", a standard of care activity to facilitate smoking cessation treatment, to patients outside of a scheduled health care appointment. The extension of this standard of care is done by offering smoking cessation coaching via MyChart instead of through providers during medical visits. Developing approaches that systematically offer treatment to all patients enrolled in the patient portal addresses several barriers identified by providers including time, lack of expertise, and concerns about the patient provider relationship. Further, it helps to increase health equity because numerous studies have demonstrated that providers are less likely to assist low-income and racial/ethnic minorities with smoking cessation treatment.

Mile Square Health Center (MSHC) has six adult primary care clinics. We will send portal messages to up to N=3000 patients randomly selected from all patients who meet eligibility criteria. Eligibility criteria includes: 1) Had an appointment at one of six MSHC (Main, Englewood, South Shore, Auburn Gresham, Cicero, Back of the Yards) clinics within the past 3 months, 2) English speaking, 3) age 18 years and older, 4) enrolled in MyChart patient portal, and 5) documented as current smoker in Epic.

The over-arching research question is: Does message (Advise) and referral approach (Refer) influence a patient's willingness to "opt-in" to receive a call from an Illinois Tobacco Quitline (ITQL) smoking cessation coach. To answer this question, patients will be randomly assigned to one of three message types delivered via the patient portal:

1. Arm 1 (Choice + Facilitated Referral): Provider advises patient to either cut down or quit smoking as a treatment goal and offers assistance in linking the patient to the ITQL. Patients indicate their acceptance of assistance by clicking the "opt-in" option to receive a call from the ITQL.
2. Arm 2 (Quit only + Facilitated Referral): Provider advises patient to quit smoking as a treatment goal and offers assistance in linking the patient to the ITQL. Patients indicate their acceptance of assistance by clicking the "opt-in" option to receive a call from the ITQL.
3. Arm 3 (Information only + Self-Referral): Provider does not advise patient to change their smoking. The Epic delivered message provides Information about the ITQL and the ITQL's telephone number to call if the patient is interested in treatment. This arm replicates the current clinic standard of care practice at MSHC because the information being provided to patients is the same, but the mode of delivery is different.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years and older
* current smoker
* English speaking
* Patient at Mile Square Health Center (Main, Englewood, South Shore, Auburn Gresham, Cicero, Back of the Yards)

Exclusion Criteria:

* aged less than 18
* non-smoker
* non English speaking
* Not a patient at MSHC

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Received Treatment | 7 months
  Number of participants who received smoking cessation counseling

SECONDARY OUTCOMES:
Smoking Cessation | 7 months
  Number of participants who quit smoking

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Caskey, MD, MaPP, Principal Investigator — University of Illinois Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Matthews AK, Watson KS, Duang C, Steffen A, Winn R. A Study Protocol for Increasing Access to Smoking Cessation Treatments for Low-Income Minority Smokers. Front Public Health. 2021 Dec 2;9:762784. doi: 10.3389/fpubh.2021.762784. eCollection 2021. PMID 34926386